CLINICAL TRIAL: NCT06989203
Title: An Intervention Study Investigating Effect of Dietary Protein Supplementation on Body Weight and Metabolic Homeostasis
Brief Title: Protein Supplementation Intervention on Body Weight
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIAS-PSITBW-202504
Record Dates: First submitted 2025-05-06; First posted 2025-05-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Weight Loss; Protein Supplementation
MeSH Terms: conditions — Obesity; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CRD (Placebo Comparator): They will receive calorie restricted balanced diet and placebo
  Interventions: Behavioral: Calorie-restricted balanced diet
- CRD+GLP-1RA (Active Comparator): They will receive calorie restricted balanced diet and semaglutide
  Interventions: Behavioral: Calorie-restricted balanced diet; Drug: semaglutide
- CRD+GLP-1RA+HP (Experimental): They will receive calorie restricted balanced diet, semaglutide, and 30g/day of dietary protein supplementation
  Interventions: Behavioral: Calorie-restricted balanced diet; Drug: semaglutide; Dietary Supplement: Dietary protein supplementation
- Healthy Comparators (Other): They will receive general lifestyle and nutritional education.
  Interventions: Behavioral: General lifestyle and nutritional education

INTERVENTIONS:
Behavioral: General lifestyle and nutritional education — Participants will receive dietary advice, behavior guidance and nutritional and lifestyle education based on dietary guidelines.
  Arms: Healthy Comparators
Behavioral: Calorie-restricted balanced diet — Participants will receive dietary advice, behavior guidance and nutritional and lifestyle education by dietitian and physicians. APP-connected wearable devices will be utilized to monitor their dietary intakes and APP-connected scale will be used to monitor their weight changes during interventions.
  Arms: CRD; CRD+GLP-1RA; CRD+GLP-1RA+HP
Drug: semaglutide — Participants will receive semaglutide as medically prescribed
  Arms: CRD+GLP-1RA; CRD+GLP-1RA+HP
Dietary Supplement: Dietary protein supplementation — participants will receive 30 g/day of dietary protein supplementation
  Arms: CRD+GLP-1RA+HP

SUMMARY:
This study is a randomized clinical trail with a parallel design, involving 120 overweight/obese (body-mass index, BMI ≥ 24 kg/m²) participants and 20 normal-weight participants. Overweight/obese participants will be randomly allocated to one of three groups: 1) calorie restricted balanced diet (CRD)group; 2) CRD + semaglutide group; or 3) CRD + segaglutide with protein supplementation. Through a 3-month weight loss intervention and 6-month follow-up, this study aims to investigate the effects of dietary protein supplementation combined with semaglutide on weight loss, energy and glucose and lipid metabolism, muscle loss, and weight regain. Additionally, the study will explore key factors affecting intervention efficacy, including obesity phenotypes, gut microbiota profiles, genetic backgrounds, and lifestyle factors, to provide evidence for optimizing individualized intervention strategies.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether adding dietary protein supplementation to GLP 1 receptor agonist (GLP-1RA, semaglutide) therapy enhances weight loss efficacy, improves energy and glucose-lipid metabolism, mitigates muscle loss, and prevents weight regain. Investigators will also explore key modifiers of treatment response-including obesity phenotype, gut microbiota composition, genetic background, and lifestyle factors-to provide an evidence base for personalized interventions.

Investigators will enroll 120 adults with overweight or obesity (BMI ≥ 24 kg/m²) and randomly assign them (1 : 1 : 1) to one of three 3 month interventions:

1. CRD: calorie restricted balanced diet;
2. CRD + GLP-1RA: CRD plus semaglutide;
3. CRD + GLP-1RA + HP: CRD plus semaglutide and 30 g/day of dietary protein supplement.

Baseline and post intervention assessments will include questionnaires; evaluations of diet, physical activity, and sleep patterns; physical examination (height, weight, waist and hip circumference, blood pressure, pulse); body composition analysis; hepatic fat and fibrosis imaging; facial skin phenotyping; 14 day continuous glucose monitoring; 14 day accelerometer based sleep and activity monitoring; stool and urine collection; and a mixed-macronutrient tolerance test (MMTT) performed in a metabolic chamber.

During the MMTT, participants consume a standardized beverage containing 126.5 g glucose, 30.67 g fat, and 34.5 g protein. Blood samples are collected at 0, 0.5, 1, 2, 3, 4, and 5 hours to characterize post prandial dynamics of energy metabolism, routine clinical biomarkers, and metabolomic profiles. Throughout the intervention, dietary intake is recorded via a mobile application, and body weight changes are tracked with an application linked smart scale.

Six months after the intervention, participants undergo follow up assessments (identical questionnaires, physical examination, fasting laboratory tests for glucose, insulin, HbA1c, lipids, and liver and renal function indices) and provide a stool sample.

To provide a healthy reference, Investigators will additionally recruit 20 normal weight adults who will receive weight maintenance dietary counseling for 3 months and undergo pre and post intervention MMTTs in the metabolic chamber. These data will help determine whether the metabolic homeostasis of overweight/obese participants after the three interventions approaches that of healthy individuals and will aid in identifying determinants of inter individual variability.

The study protocol has been approved by the Ethics Committee of Zhejiang Provincial Tongde Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 50 years.
* Normal-weight participants: 18.5 kg/m² ≤ Body Mass Index (BMI) < 24 kg/m².
* Overweight or obese participants:

BMI ≥ 28 kg/m², or 24 kg/m² ≤ BMI < 28 kg/m² and a clinical diagnosis meeting semaglutide treatment indications (e.g., hyperglycemia, hypertension, dyslipidemia, fatty liver, obstructive sleep apnea, cardiovascular disease, etc.).

* Willingness to participate in this study and provide signed informed consent.

Exclusion Criteria:

* Abnormal metabolic indicators (meeting any one of the following criteria is grounds for exclusion):

  1. Normal weight (18.5 kg/m² ≤ BMI < 24 kg/m²):
  1. Waist circumference ≥ 90 cm for men or ≥ 85 cm for women.
  2. Fasting glucose ≥ 6.1 mmol/L or 2-hour postprandial glucose ≥ 7.8 mmol/L, or a confirmed diagnosis of diabetes.
  3. Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg, or currently under antihypertensive treatment.
  4. Fasting triglycerides (TG) ≥ 1.7 mmol/L; high-density lipoprotein cholesterol (HDL-C) < 0.9 mmol/L in men or < 1.0 mmol/L in women.

  2. Overweight or obese (BMI ≥ 24 kg/m²):
  1. Fasting plasma glucose > 11.1 mmol/L or HbA1c > 9%, or previously diagnosed diabetes, or currently using insulin or any antidiabetic medication.
  2. Blood pressure ≥ 160/100 mmHg, or clinically diagnosed stage 2 or stage 3 (moderate or severe) hypertension, or currently under antihypertensive treatment.
  3. Use of lipid-lowering drugs (e.g., fibrates, bile acid sequestrants, statins, PCSK9 inhibitors) within the past 3 months, or TG ≥ 5.7 mmol/L, or LDL ≥ 4.9 mmol/L.
* Pregnancy or lactation.
* Self-reported weight change of more than 5 kg within the 90 days prior to screening.
* Use of antibiotics, antimicrobials, or anti-inflammatory/analgesic salicylates (e.g., aspirin) within the 3 months prior to screening for 3 days or more.
* Use of estrogen therapy or other hormonal medications within the past 6 months.
* Use of GLP-1 receptor agonists or probiotics within the past 3 months.
* Heavy alcohol consumption (females > 40 g/day, approximately 250 mL of huangjiu [yellow rice wine], or 1000 mL of beer, or 100 mL of liquor per day; males > 80 g/day).
* Severe liver or kidney dysfunction (ALT, AST, or serum creatinine exceeding 3 times the upper limit of normal, UACR ≥ 30 mg/g, or eGFR < 60 mL/min).
* Gastrointestinal diseases affecting digestion and absorption (e.g., severe diarrhea, severe constipation, severe inflammatory bowel disease, peptic ulcer, gallstones, cholecystitis).
* Underwent surgery within the past year (excluding appendectomy or hernia repair).
* Severe cardiovascular or cerebrovascular diseases (e.g., heart failure, myocardial infarction, stroke, acute myocarditis, severe arrhythmia, or receiving interventional therapy).
* Presence of metallic implants such as a cardiac stent or pacemaker.
* Cancer or having received radiation or chemotherapy within the past 5 years.
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia, or a personal history of hyperthyroidism or hypothyroidism.
* Chronic or acute pancreatitis.
* Positive hepatitis B surface antigen (HBsAg), active tuberculosis, HIV, or other infectious diseases.
* Currently participating in another clinical study or having done so within the past 3 months.
* Claustrophobia.
* Any psychiatric disorder such as attention-deficit/hyperactivity disorder (ADHD), bipolar disorder, or epilepsy (including current use of antiepileptic medications), or use of antidepressant medications.
* Inability to read, write, operate a smartphone, or perform daily activities independently.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Body Weight (kg) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Weight will be assessed using a Seca-255 scale (ScalesGalore).

SECONDARY OUTCOMES:
Change in Energy Expenditure Rate (kcal/minute) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Energy expenditure rate (kcal/minute) will be assessed with a whole-room indirect calorimeter.
Change in Respiratory Quotient from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Respiratory quotient will be assessed with a whole-room indirect calorimeter.
Change in Fat Oxidation Rate (g/minute) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Fat oxidation rate (g/minute) will be assessed with a whole-room indirect calorimeter.
Change in Carbohydrate Oxidation Rate (g/minute) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Carbohydrate oxidation rate (g/minute) will be assessed with a whole-room indirect calorimeter.
Change in Waist Circumference (cm) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Waist circumference will be assessed using a Seca-201tape (ScalesGalore).
Change in Hip Circumference (cm) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Hip circumference will be assessed using a Seca-201 tape (ScalesGalore).
Change in Fat-free Mass (kg) From Baseline to Week 12 | Baseline (Week 0) and Week 12
  Absolute change in whole-body fat-free mass measured by dual-energy X-ray absorptiometry (DXA; GE Lunar iDXA).
  Values at Week 12 will be subtracted from baseline; a positive value indicates an increase in fat-free mass.
Change in Fat Mass (kg) From Baseline to Week 12 | Baseline (Week 0) and Week 12
  Absolute change in whole-body fat mass measured by dual-energy X-ray absorptiometry (DXA; GE Lunar iDXA).
  Values at Week 12 minus baseline; a positive value indicates an increase in fat mass.
Change in Controlled Attenuation Parameter (CAP, dB/m) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. CAP will be assessed using FibroScane (Echosens). The median CAP value of 10 valid measurements will be used (IQR ≤ 30%). Reported value = Week 12 CAP minus baseline CAP; positive values indicate increased hepatic steatosis.
Change in Systolic Blood Pressure (mmHg) from Baseline to Week 12 | Baseline and Week 12
  The change in systolic blood pressure between the baseline and after 12-week intervention. Systolic blood pressure will be assessed with an electronic blood pressure monitor (Omron J750).
Change in Diastolic Blood Pressure (mmHg) from Baseline to Week 12 | Baseline and Week 12
  The change in diastolic blood pressure between the baseline and after 12-week intervention. Diastolic blood pressure will be assessed with an electronic blood pressure monitor (Omron J750).
Change in Heart Rate (beats/minute) from Baseline to Week 12 | Baseline and Week 12
  The change in heart rate between the baseline and after 12-week intervention. Heart rate will be assessed using Omron J750.
Change in Fasting Glucose (mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change of fasting glucose between the baseline and after 12-week intervention. Glucose will be measured using a hexokinase enzymatic assay.
Change in Glucose Incremental AUC (mmol·min/L) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an oral mixed-meal tolerance test (MMTT). Glucose will be measured using a hexokinase enzymatic assay. Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in HbA1c (%) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. HbA1c will be assessed using high-performance liquid chromatography
Change in Fasting Insulin (µIU/mL) from Baseline to Weel 12 | Baseline and Week 12
  The change of fasting insulin between the baseline and after 12-week intervention. Insulin will be measured using an electrochemiluminescence assay.
Change in Insulin Incremental AUC (µIU·min/mL) from Baseline to Weel 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. Insulin will be measured using an electrochemiluminescence assay. Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Fasting C-peptide (ng/mL) from Baseline to Week 12 | Baseline and Week 12
  The change of fasting C-peptide between the baseline and after 12-week intervention. C-peptide will be measured using an electrochemiluminescence assay.
Change in C-peptide Incremental AUC (ng·min/mL) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. C-peptide will be measured using an electrochemiluminescence assay. Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Mean 24-h Glucose (mg/dL) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Mean 24-h glucose will be assessed using Continuous Glucose Monitoring (FreeStyle Libre 2, Abbott) for 14 consecutive days.
Change in Glucose Coefficient of Variation (CV, %) from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week intervention. Glucose CV) will be calculated as (SD/mean) × 100 % from continuous glucose monitoring (FreeStyle Libre 2, Abbott). Participants will wear the sensor for 14 consecutive days at each time point.
Change in Fasting Serum Triglycerides (mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change of fasting serum triglycerides between the baseline and after 12-week intervention. Serum triglycerides will be quantified using an enzymatic colorimetric assay.
Change in Triglyceride Incremental AUC (mmol·min/L) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. Triglyceride will be measured using an enzymatic colorimetric assay. Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Fasting Serum Total Cholesterol (mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change of fasting total cholesterol between the baseline and after 12-week lifestyle intervention. Total cholesterol will be quantified in serum using an enzymatic colorimetric assay.
Change in Total Cholesterol Incremental AUC (mmol·min/L) from Baseline at 12 Weeks | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. Total cholesterol will be measured using an enzymatic colorimetric assay. Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Fasting Serum High-Density Lipoprotein Cholesterol (HDL-C, mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change of fasting HDL-C between the baseline and after 12-week lifestyle intervention. HDL-C will be quantified in serum using an enzymatic colorimetric assay.
Change in HDL-c Incremental AUC (mmol·min/L) from Baseline to 12 Weeks | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. HDL-c will be measured using an enzymatic colorimetric assay. Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in Fasting Serum Low-Density Lipoprotein Cholesterol (LDL-C, mmol/L) from Baseline to Week 12 | Baseline and Week 12
  The change of fasting LDL-C between the baseline and after 12-week lifestyle intervention. LDL-C will be quantified in serum using an enzymatic colorimetric assay.
Change in LDL-c Incremental AUC (mmol·min/L) from Baseline to 12 Weeks | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. LDL-c will be measured using an enzymatic colorimetric assay. Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value. Reported value = Week 12 iAUC - baseline iAUC; positive numbers indicate an increase.
Change in GLP-1 Incremental AUC (pg·min/mL) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. GLP-1 will be quantified using a high-sensitivity ELISA . Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value.
Change in GIP Incremental AUC (pg·min/mL) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. GIP will be quantified using a high-sensitivity ELISA . Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value.
Change in Ghrelin Incremental AUC (pg·min/mL) from Baseline to Week 12 | Baseline and Week 12
  Venous blood will be collected at 0, 30, 60, 120, 180, 240, and 300 min during an MMTT. Ghrelin will be quantified using a high-sensitivity ELISA . Incremental area under the concentration-time curve (iAUC) will be calculated via the trapezoidal rule after subtracting the fasting value.
Change in Shannon Diversity Index From Baseline to Week 12 | Baseline and Week 12
  Fecal DNA will be extracted and subjected to shotgun metagenomic sequencing on an Illumina NovaSeq 6000 (2 × 150 bp; ≥6 Gb per sample). Reads will be taxonomically profiled using MetaPhlAn 4.0. The Shannon diversity index will be calculated for each sample.
Change in Relative Abundance of Akkermansia muciniphila (%) From Baseline to Week 12 | Baseline and Week 12
  Same sequencing workflow as above. Relative abundance (% of total classified reads) of A. muciniphila will be extracted from MetaPhlAn output. Reported value = Week 12 minus baseline abundance.
Single nucleotide polymorphism (SNPs) | Baseline
  Mutations at specific sites will be detected using a genotyping microarray.
Change in body weight from Week 12 to 6 months post-intervention | Post-intervention 6 months
  The hange from the end of intervention (Week 12) to 6 months post-intervention. Weight will be assessed using Seca-255 scale (ScalesGalore).
Change in Facial Skin Phenotype from Baseline to Week 12 | Baseline and Week 12
  The change between the baseline and after 12-week lifestyle intervention.Facial skin phenotype will assessed using Meitueve 3D skin analysis system (Meitu, China).

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, PhD, Principal Investigator — Institute for Nutritional Sciecnes, CAS; Hangzhou Institute for Advanced Study, UCAS
Locations (1):
- Hangzhou Institute for Advanced Study, University of Chinese Academy of Sciences, Hangzhou, Zhejiang, China